CLINICAL TRIAL: NCT05620056
Title: A Population-based Study of Drug Exposures and Adverse Pregnancy Outcomes in China (DEEP)
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: Xiamen Health Commission (Unknown); Xiamen Health and Medical Big Data Center (Unknown)
Responsible Party: Principal Investigator, Sun Xin, Director of Chinese Evidence-based Medicine Center, West China Hospital
Other Study IDs: DEEP
Record Dates: First submitted 2022-11-03; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy; Congenital Malformation; Drug Exposure
Keywords: Cohort study; drug exposures; congenital malformation; pregnancy; population-based
MeSH Terms: conditions — Congenital Abnormalities | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- drug exposure: chemicals drugs, biological products, patent Chinese Medicines, Chinese herbs
  Interventions: Drug: chemicals drugs, biological products, patent Chinese Medicines, Chinese herbs

INTERVENTIONS:
Drug: chemicals drugs, biological products, patent Chinese Medicines, Chinese herbs — medication (i.e., chemicals drugs, biological products, patent Chinese Medicines, Chinese herbs ) exposure through the pregnancy life course

SUMMARY:
The DEEP cohort is the first population-based cohort of pregnant population in China that longitudinally documents drug uses throughout the pregnancy life course and adverse pregnancy outcomes.

DETAILED DESCRIPTION:
The DEEP cohort is the first population-based cohort of pregnant population in China that longitudinally documents drug uses throughout the pregnancy life course and adverse pregnancy outcomes. The main goal of the study aims to monitor and evaluate the safety of drug use through the pregnancy life course in the Chinese setting. The DEEP cohort is developed primarily based on the population-based data platforms in Xiamen, a municipal city of 5 million population in southeast China. Based on these data platforms, a pregnancy-centered registry was developed that documented health care services and outcomes in the maternal and other departments. For identifying drug uses, a drug prescription database was specifically developed by using electronic healthcare records documented in the platforms across the primary, secondary and tertiary hospitals. By linking the pregnancy registry and prescription database through a unique identifier, the DEEP cohort was developed. All the pregnant women and their offspring in Xiamen are provided with health care and followed up according to standard protocols in the region, including antenatal care, delivery care, postpartum follow-up and childhood follow-ups. The primary adverse outcomes - congenital malformations - are collected using a standardized Case Report Form.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who registered at the Maternal and Child Health Management Platform in Xiamen.

Exclusion Criteria:

* None

Ages: 14 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All pregnant women registered at the Maternal and Child Health Management Platform were enrolled.
Study Population: From January 2013, all pregnant women who registered at the Maternal and Child Health Management in Xiamen was included in this cohort.
Sampling Method: Probability Sample
Enrollment: 564760 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
congenital malformations | up to 42 days after delivery
  Number of births with congenital malformations

SECONDARY OUTCOMES:
preterm birth | up to 37 gestational weeks
  Number of pregnancies with preterm birth
low birth weight | Immediately after delivery
  Number of live births with low birth weight

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, Study Chair — Chinese Evidence-based Medicine Center, West China Hospital, Sichuan University, Chengdu, 610041, China
Locations (1):
- Xiamen Health and Medical Big Data Center, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Following the policy of Xiamen Health Commission, research institutions could apply for data access by submitting a formal study protocol, subjected to approval by the Xiamen Health and Medical Big Data Center and the Chinese Evidence-based Medicine Center. Ethical review and research registration are mandatory for all studies.
Supporting Information: Study Protocol, SAP